CLINICAL TRIAL: NCT03156751
Title: Feasibility of Introducing an Onsite Test for Syphilis in the Package of Antenatal Care at the Rural Primary Health Care Level in Burkina Faso
Brief Title: Feasibility of Introducing an Onsite Test for Syphilis in the Package of Antenatal Care in Burkina Faso
Status: Completed | Type: Observational
Sponsor: Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government)
Collaborators: World Health Organization (Other); African Population and Health Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: IRSS003
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Syphilis Infection; Diagnoses Disease
Keywords: Syphilis screening; antenatal care; prenatal diagnosis; rapid diagnosis test; Burkina Faso; feasibility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Feasibility of introducing onsite test for syphilis in the package of antenatal care at rural primary health care in Burkina Faso — This study used a pre post intervention mixed methods quasi-experimental design with a group of health facilities offering ANC services. It was conducted in three phases, which consisted of a situational analysis using qualitative methods (Phase 1), selecting an appropriate test through evaluating 4 candidate tests and the participatory design and implementation of an intervention(Phase 2), and an evaluation combining review of record tools, interviews, time motion study and estimating incremental costs (Phase 3). The conceptual framework draws on multilevel assessment (MLA), policy triangle framework, MRC framework for designing complex interventions and the Normalization Process Model (NPM). The findings suggested that an intervention that introduces point of care test for syphilis at antenatal care services is feasible, acceptable, and of comparable costs to HIV screening in pregnancy. Nonetheless, barriers identified by health workers need to be overcome.

SUMMARY:
This study used a pre post intervention mixed methods quasi-experimental design with a group of health facilities offering antenatal care (ANC) services (primary health centers in rural area) as the sampling units. This study was conducted in three phases, which consisted of a situational analysis using qualitative methods (Phase 1), selecting an appropriate test through evaluating 4 candidate tests and the participatory design and implementation of an intervention that included onsite training, provision of supplies and medicines, quality control and supervision (Phase 2), and an evaluation combining review of record tools, interviews, time motion study and estimating incremental costs (Phase 3). The conceptual framework draws on multilevel assessment (MLA), policy triangle framework, Medical Research Council framework for designing complex interventions and the Normalization Process Model (NPM). Methods included document review, seventy five interviews were conducted with health providers, district managers, facility managers, traditional healers, pregnant women, community health workers, and Non-Governmental Organizations (NGO) managers in phase I and fourteen in phase III, non-participant observation, time-motion study, incremental cost analysis, and sensitivity, specificity and ease of use analysis of four candidate point-of care tests. Data were collected between 2012 and 2014. Qualitative data were analyzed through thematic analysis supported by Nvivo software. Quantitative data were analyzed through descriptive statistics such as frequency, mean and median supported by SPSS. Phase I identified barriers to implementation and uptake of syphilis testing at health provider and community levels. The most important barriers at provider level included fragmentation of services, poor communication between health workers and clients, failure to prescribe syphilis test, and low awareness of syphilis burden. Cost of testing, distance to laboratory and lack of knowledge about syphilis were identified as barriers at community level. Phase II: Alere DetermineTM Syphilis was the most sensitive of the four point-of-care tests evaluated. The components of the intervention were successfully implemented in the selected health facilities. Overall, phase III showed that it is feasible and acceptable to introduce a point of care test for syphilis in antenatal care services at primary health care level using the available staff. The findings suggested that an intervention that introduces point of care test for syphilis at antenatal care services is feasible, acceptable, and of comparable costs to HIV screening in pregnancy. Nonetheless, instructions and supervision need to be clearer to achieve optimal levels of screening and quality control, and barriers identified by health workers need to be overcome. The point-of care test for syphilis is likely to be acceptable by health workers as a routine service and incorporated as a normal practice in Burkina Faso context.

ELIGIBILITY:
Inclusion Criteria:

* pregnant woman aged 18 and over at first antenatal care visit
* pregnant woman who gave consent for receiving rapid diagnosis test

Exclusion Criteria:

* Pregnant woman aged less than 18 years
* Pregnant woman not at their first antenatal care visit
* Pregnant woman who did not give her consent for receiving rapid diagnosis test

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women coming for antenatal care visit at selected health facilities in Kaya health district
Sampling Method: Non-Probability Sample
Enrollment: 1205 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2013-09-30 (Actual); Study Completion 2013-09-30 (Actual)

PRIMARY OUTCOMES:
Pregnant women who were screened for syphilis | may 2013 to september 2013
  Number of pregnant women who received rapid diagnostic test for syphilis

CONTACTS AND LOCATIONS:
Overall Officials: Seni KOUANDA, PhD, Principal Investigator — Insitut de Recherche en Science de la santé; Fadima YAYA BOCOUM, PhD, Study Director — Insitut de Recherche en Science de la santé

IPD SHARING:
Plan to Share IPD: No
The individual participant data could be obtained if requested by other researchers to the principal investigator.

REFERENCES:
- [Derived] Bocoum FY, Tarnagda G, Bationo F, Savadogo JR, Nacro S, Kouanda S, Zarowsky C. Introducing onsite antenatal syphilis screening in Burkina Faso: implementation and evaluation of a feasibility intervention tailored to a local context. BMC Health Serv Res. 2017 May 30;17(1):378. doi: 10.1186/s12913-017-2325-x. PMID 28558812